CLINICAL TRIAL: NCT01017783
Title: Randomized Controlled Trial of a Water Beverage Intervention for Promoting Modest Weight Reduction in Free Living Adults
Brief Title: Trial of a Water Beverage Intervention for Promoting Modest Weight Reduction in Free Living Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Nestle Waters North America, Inc (Unknown)
Responsible Party: Deborah F. Tate, PhD, The University of North Carolina at Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNC-Nestle-01
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy Choices (Other)
  Interventions: Behavioral: Healthy Choices
- Diet Substitution A (Experimental)
  Interventions: Behavioral: Dietary substitution A
- Diet Substitution B (Experimental)
  Interventions: Behavioral: Dietary Substitution B

INTERVENTIONS:
Behavioral: Dietary substitution A — Substitution of calorie-dense item with lower calorie choice A
  Arms: Diet Substitution A
Behavioral: Dietary Substitution B — Substitution of calorie-dense item with lower calorie option B
  Arms: Diet Substitution B
Behavioral: Healthy Choices — Multiple healthy choices presented with self-selection of choices used
  Arms: Healthy Choices

SUMMARY:
The primary objectives of this clinical trial are to determine if replacing sugar sweetened beverages with water consumption promote weight loss over 6 months in overweight adults and if replacing sugar sweetened beverages with water consumption promote greater weight loss over 6 months relative to replacement with other non-caloric sweetened beverages or control.

The secondary objective is to identify mediators and moderators of the effect of water replacement including hydration status, glucose metabolism, anthropometrics, physical activity, dietary intake and resting metabolic rate.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age.
* Body mass index (BMI) between 25.0-49.9 kg/m2.
* Subject consumes at least 280 calories per day from caloric beverages.

Exclusion Criteria:

* Report losing >5% of current body weight in the previous 6 months.
* Report participating in a research project involving weight loss or physical activity in the previous 6 months, as these proximal experiences may impact the results of this study. Additionally, report current participating in any other research studies whose results could be compromised by or in which participation could compromise this research study. (Participation in a research study that would not affect or be affected by this study is allowed.)
* Report pregnancy or lactation during the previous 6 months, or planned pregnancy in the next 6 months.
* Report taking medication that could affect metabolism or change body weight (e.g., synthroid).
* Report hospitalization for psychiatric problems during the prior year.
* Report major psychiatric diagnoses and organic brain syndromes.
* Report heart problems, chest pain, cancer within the last 5 years
* Being treated by a therapist for psychological issues or problems with psychotropic medications.
* Report behaviors that indicate probable alcohol dependence as assessed by the Rapid Alcohol Problems Screen (RAPS4-QF) (Cherpitel CJ, 2002).
* Unwilling to change intake of beverages during the study period.
* Plan to move from the area during the study period, and/or unable to attend monthly group meetings.
* Report not having adequate transportation to the study center that would allow transport of study supplies back to the subject's home.
* Report not being able to attend group meetings on Monday or Tuesday evenings.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Weight change | 0, 3, 6 months

SECONDARY OUTCOMES:
urine specific gravity | 0, 3, 6 months
fasting glucose | 0, 3, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Deborah F Tate, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Piernas C, Tate DF, Wang X, Popkin BM. Does diet-beverage intake affect dietary consumption patterns? Results from the Choose Healthy Options Consciously Everyday (CHOICE) randomized clinical trial. Am J Clin Nutr. 2013 Mar;97(3):604-11. doi: 10.3945/ajcn.112.048405. Epub 2013 Jan 30. PMID 23364015
- [Derived] Tate DF, Turner-McGrievy G, Lyons E, Stevens J, Erickson K, Polzien K, Diamond M, Wang X, Popkin B. Replacing caloric beverages with water or diet beverages for weight loss in adults: main results of the Choose Healthy Options Consciously Everyday (CHOICE) randomized clinical trial. Am J Clin Nutr. 2012 Mar;95(3):555-63. doi: 10.3945/ajcn.111.026278. Epub 2012 Feb 1. PMID 22301929